CLINICAL TRIAL: NCT02405234
Title: Safety and Effectiveness Study of Ascension PyroCarbon Radial Head Compared to Ascension Metal Radial Head
Brief Title: Ascension PyroCarbon Radial Head Study
Acronym: CMRH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-RH-002; NCT00825409 (obsolete NCT alias)
Record Dates: First submitted 2014-11-04; First posted 2015-04-01 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2017-08

CONDITIONS: Degenerative Arthritis; Radial Head Fracture; Rheumatoid Arthritis
Keywords: Radial Head Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Radial Head and Neck Fractures; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Carbon Modular Radial Head (Experimental): PyroCarbon Modular Radial Head replacement
  Interventions: Device: Carbon Modular Radial Head replacement
- Metal Radial Head (Active Comparator): Metal Radial Head replacement
  Interventions: Device: Metal Radial Head replacement

INTERVENTIONS:
Device: Carbon Modular Radial Head replacement — 'Carbon Modular Radial Head replacement: The Ascension Radial Head is made of pyrocarbon, a material that testing has shown to be both wear resistant and biocompatible and has been used in surgical implants for years. The introduction of the pyrocarbon head should alleviate the problems associated with wear debris and fragmentation experienced with the silicone radial spacer.
  Other Names: Ascension CMRH
  Arms: Carbon Modular Radial Head
Device: Metal Radial Head replacement — Metal Radial Head replacement:The Ascension® Modular Radial Head (MRH) is an anatomically designed, single-use, modular prosthesis designed for replacement of the proximal end of the radius. FDA cleared this device for commercial distribution under 510(k) K032686. It is made from medical grade cobalt chromium alloy meeting ASTM F1537. Head components are available in six sizes and stem components are available in four sizes are interchangeable and assembled with a taper connection.
  Other Names: Ascension MRH
  Arms: Metal Radial Head

SUMMARY:
The proportion of patient successes with the Carbon Modular Radial Head at the 2-year evaluation is no lower than the proportion of patient successes with the Metal Radial Head.

DETAILED DESCRIPTION:
This investigation will include 179 patients (119 study devices and 60 control devices) enrolled at 15 active centers. In addition a subset of 24 RA patients will be enrolled and analyzed separately. The trial is designed as a randomized, non-inferiority study comparing results of the CMRH to results of the MRH.

This will be a multi-site study with all patients either receiving the CMRH or the MRH. Sequential enrollment of all patients meeting inclusion criteria and agreeing to be in the study will be enrolled. The patients will sign an informed consent agreeing to accept either the investigational or control device. In addition, the surgeon will not know which device the patient is to receive until the day of surgery in an attempt to further reduce bias. The surgeon will open an envelope at the time of surgery to determine if a CMRH or MRH will be implanted.

Additional efforts to eliminate bias in the study will include a final radiographic analysis by an independent observer experienced in reporting on orthopedic devices. The independent reviewer will grade the surgical implant and determine radiographic success/failure for each patient.

Implants will be assigned to patients at the clinical sites in a block randomization fashion. The randomization will be site specific. At a given site, each consecutive block of six enrolled patients to be treated will receive random assignments of CMRH or MRH at a 2:1. The randomization schedule is generated by computer (NQuery) and is produced in blocks of 6, where 4 are study devices and 2 are control devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients must need a radial head replacement for:

  * Degenerative, post-traumatic or rheumatoid arthritis
  * Primary replacement after fracture of the radial head
  * Relief of symptoms after radial head resection
  * Revision of failed radial head arthroplasty
  * Skeletally mature individuals ages 18 - 85

Exclusion Criteria:

* Inadequate bone stock or soft tissue coverage
* Previous open fracture or infection in the joint
* Individuals under age of 18 or over 85 years of age
* Physical interference with or by other prostheses during implantation or use
* Procedures requiring modification of the prosthesis
* Skin, bone, circulatory and/or neurological deficiency at the implantation site
* Prisoners
* Patients on chronic corticosteroid or non-steroidal anti-inflammatory therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2015-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patient successes with the Carbon Modular Radial Head vs patient successes with the Metal Radial Head as assessed by implant survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tummon, Study Director — Integra Life Sciences
Locations (4):
- United States (4):
  - University of Florida Orthopedic and Rehabilitation, Gainesville, Florida
  - Hand Center of Southwestern Ohio, Dayton, Ohio
  - The Rothman Institute, Philadelphia, Pennsylvania
  - Texas Orthopedic Hospital, Houston, Texas